CLINICAL TRIAL: NCT04046237
Title: Impact of Treating Severe Periodontitis on Inflammatory Activity of Atheromatous Plaques in Patients With Acute Myocardial Infarction (AMI)
Acronym: PAROCARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P171104
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Acute Myocardial Infarction; Severe Periodontitis; Carotid Atherosclerosis
Keywords: Acute Myocardial Infarction; Severe Periodontitis; FDG-PET; Carotid Atherosclerosis
MeSH Terms: conditions — Periodontitis; Carotid Artery Diseases | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual treatment - Control group (No Intervention): The patient is referred to his treating dentist with a diagnosis report of his oral state including his periodontal status.
  The usual care usually includes the extraction of non-preservable teeth, the dental prosthesis to replace them and at least one descaling session.
- Periodontal treatment - Intervention group (Experimental): Periodontal treatment can last up to 6 months depending on the periodontal state, followed by a follow-up period of at least 6 months including a visit at M9.
  Briefly, the intervention group includes initial therapy with information on oral hygiene techniques, scaling and surfacing of dental roots. This initial therapy is followed by a resumption of periodontal clinical measures after 6 weeks. Depending on the degree of improvement of the measurements, the treatment is either completed, or continues with further scaling-surfacing and / or performing one or more periodontal surgeries. Periodontal monitoring period often called "maintenance" includes repeated sessions of simple scaling whose rate does not exceed 4 per year.
  Interventions: Other: Periodontal treatment

INTERVENTIONS:
Other: Periodontal treatment — Periodontal treatment can last up to 6 months depending on the periodontal state, followed by a follow-up period of at least 6 months including a visit to M9.
  Briefly, the intervention group includes initial therapy in 48 hours maximum which includes information on oral hygiene techniques (verbal + brochure), scaling and surfacing of dental roots with antiseptic irrigation and non-tooth extraction. retainable. This initial therapy is followed by a resumption of periodontal clinical measures after 6 weeks. Depending on the degree of improvement of the measurements, the treatment is either completed, or continues with further scaling-surfacing and / or performing one or more periodontal surgeries. Periodontal monitoring period often called "maintenance" includes repeated sessions of simple scaling whose rate does not exceed 4 per year.
  Arms: Periodontal treatment - Intervention group

SUMMARY:
Multicenter randomized clinical trial with two arms in patients hospitalized for an AMI nested in the Frenchie registry. Periodontal therapy is performed by periodontists in the intervention group versus treatment by dental surgeons as part of their usual practice in the control group.

For the intervention group, periodontal management will be carried out for a maximum of 6 months after randomisation, prolonged by a follow-up of 6 months including a maintenance visit at M9.

All patients will have an FDG-PET at M0 and M12 for evaluation of inflammation on carotid atherosclerotic plaques.

DETAILED DESCRIPTION:
Eligible adults 30 to 70 years old hospitalized for an MI, (cf inclusion and non-inclusion criteria), will be asked to participate in the study. (screening)

At M0 :

* patients will be examined by a periodontist for assessing the severity of periodontitis (standard oral examination including a periodontal screening test).
* Patients with severe periodontitis will then receive: Complete periodontal examination of all teeth (6 sites per tooth) including pocket depth measurement, measurement of gingival recession, plaque index, gingival bleeding index, and a gingival fluid sample. Patients will then be informed of their periodontal status and therapeutic options. At this point, the patient may decide not to follow the treatment and will not be randomized.
* Patients who agree to continue the study will have a venous blood sample and a PET-FDG examination. Patients in whom the acquisition of FDG-PET is impossible will not be randomized.

At the end of these examinations, if all the conditions are met, the randomization will be carried out :

* Intervention group: Periodontal treatment, for a maximum of 6 months. At the end of the periodontal treatment, a follow-up of at least 6 months, including a maintenance visit to M9, will be performed.
* Control group: patients will be referred to their treating dentist for usual care.

At M12 (+12 months) : All patients (intervention group and control group) will have the same tests as M0

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for an acute myocardial infarction and included in the Frenchie registry
* Score ≥ 5 on the screening questionnaire for periodontitis
* Six teeth at least (excluding wisdom teeth)
* Consent signature
* Affiliation to a French medical insurance (Sécurité Sociale)

Exclusion Criteria:

* Patients with diseases,other than cardiovascular and diabetes, known to change the periodontal state such as AIDS, rheumatoid arthritis, Chediak-Higashi syndrome, Papillon-Lefèvre
* Systemic antibiotic therapy> 48 hours in the 3 months prior to inclusion
* Acute heart failure
* Uncontrolled ventricular rhythm disorders
* Impossibility for the patient to attend follow-up visits
* Impossibility to maintain the extended position for 20 minutes
* Immunosuppressive therapy> 1 month in the 6 months prior to inclusion
* Pregnancy, breastfeeding
* Known hypersensitivity to chlorhexidine, povidone, 18-fluoro-deoxyglucose

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Effect of treatment of severe periodontitis in patients with an AMI | 12 months (+12months) after randomization
  The primary endpoint will be the absolute difference of the Most-Diseased Segment (MDS) -Target to Background Ratio (TBR) measured at the segment with the highest activity on carotid arteries between the initial PET scan and the PET scan performed at 12 months (+12months) after randomization

SECONDARY OUTCOMES:
Effect of treatment of severe periodontitis in patients with an AMI | 12 months (+12months) after randomization
  Relative difference of the most-diseased segment (MDS) Tissue to Background ratio (TBR) ((M12-M0)/M0) of the Most-Diseased Segment (MDS) -Target to Background Ratio (TBR) measured at the segment with the highest activity
Impact of periodontitis treatment on the intensity of global inflammatory activity measured in the alveolar bone | 12 months (+12months) after randomization
  Relative ((M12-M0)/M0) and absolute (M12-M0) differences of TBR in the alveolar bone
Impact of periodontitis treatment on the intensity of global inflammatory activity measured in the thoracic aorta | 12 months (+12months) after randomization
  Relative ((M12-M0)/M0) and absolute (M12-M0) differences of mean TBR in the thoracic aorta
Dysbiosis | 12 months (+12months) after randomization
  Changes in the dysbiosis index
CD31 in plasma and gingival fluid | 12 months (+12months) after randomization
  Changes in concentrations of soluble CD31 in plasma and the gingival fluid
Inflammatory markers concentrations in the gingival fluid and in the plasma | 12 months (+12months) after randomization
  Changes in the inflammatory markers including IL-1β, IL-6, IL-8, TNFalpha, MMP8, MMP9 concentrations in the gingival fluid and in the plasma
Evaluation of overall inflammation in vascular arteries | At randomization
  Correlation between soluble CD31 / cleaved CD31 ratio and TBR
Evaluation of TBR measurments according to glycemia values | 12 months (+12months) after randomization
  Evaluation of TBR measurments according to glycemia values measured prior to FDG-PET

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gabriel STEG, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lockhart PB, Bolger AF, Papapanou PN, Osinbowale O, Trevisan M, Levison ME, Taubert KA, Newburger JW, Gornik HL, Gewitz MH, Wilson WR, Smith SC Jr, Baddour LM; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee of the Council on Cardiovascular Disease in the Young, Council on Epidemiology and Prevention, Council on Peripheral Vascular Disease, and Council on Clinical Cardiology. Periodontal disease and atherosclerotic vascular disease: does the evidence support an independent association?: a scientific statement from the American Heart Association. Circulation. 2012 May 22;125(20):2520-44. doi: 10.1161/CIR.0b013e31825719f3. Epub 2012 Apr 18. PMID 22514251
- [Background] Tonetti MS, Van Dyke TE; working group 1 of the joint EFP/AAP workshop. Periodontitis and atherosclerotic cardiovascular disease: consensus report of the Joint EFP/AAP Workshop on Periodontitis and Systemic Diseases. J Periodontol. 2013 Apr;84(4 Suppl):S24-9. doi: 10.1902/jop.2013.1340019. PMID 23631582
- [Background] LaMonte MJ, Genco RJ, Hovey KM, Wallace RB, Freudenheim JL, Michaud DS, Mai X, Tinker LF, Salazar CR, Andrews CA, Li W, Eaton CB, Martin LW, Wactawski-Wende J. History of Periodontitis Diagnosis and Edentulism as Predictors of Cardiovascular Disease, Stroke, and Mortality in Postmenopausal Women. J Am Heart Assoc. 2017 Mar 29;6(4):e004518. doi: 10.1161/JAHA.116.004518. PMID 28356279
- [Background] Adolph M, Darnaud C, Thomas F, Pannier B, Danchin N, Batty GD, Bouchard P. Oral health in relation to all-cause mortality: the IPC cohort study. Sci Rep. 2017 Mar 15;7:44604. doi: 10.1038/srep44604. PMID 28294149
- [Background] Schmitt A, Carra MC, Boutouyrie P, Bouchard P. Periodontitis and arterial stiffness: a systematic review and meta-analysis. J Clin Periodontol. 2015 Nov;42(11):977-87. doi: 10.1111/jcpe.12467. Epub 2015 Nov 24. PMID 26465940
- [Background] Piconi S, Trabattoni D, Luraghi C, Perilli E, Borelli M, Pacei M, Rizzardini G, Lattuada A, Bray DH, Catalano M, Sparaco A, Clerici M. Treatment of periodontal disease results in improvements in endothelial dysfunction and reduction of the carotid intima-media thickness. FASEB J. 2009 Apr;23(4):1196-204. doi: 10.1096/fj.08-119578. Epub 2008 Dec 12. PMID 19074511
- [Background] Tonetti MS, D'Aiuto F, Nibali L, Donald A, Storry C, Parkar M, Suvan J, Hingorani AD, Vallance P, Deanfield J. Treatment of periodontitis and endothelial function. N Engl J Med. 2007 Mar 1;356(9):911-20. doi: 10.1056/NEJMoa063186. PMID 17329698
- [Background] Hajishengallis G. Periodontitis: from microbial immune subversion to systemic inflammation. Nat Rev Immunol. 2015 Jan;15(1):30-44. doi: 10.1038/nri3785. PMID 25534621
- [Background] Eke PI, Dye BA, Wei L, Slade GD, Thornton-Evans GO, Borgnakke WS, Taylor GW, Page RC, Beck JD, Genco RJ. Update on Prevalence of Periodontitis in Adults in the United States: NHANES 2009 to 2012. J Periodontol. 2015 May;86(5):611-22. doi: 10.1902/jop.2015.140520. Epub 2015 Feb 17. PMID 25688694
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Bahekar AA, Singh S, Saha S, Molnar J, Arora R. The prevalence and incidence of coronary heart disease is significantly increased in periodontitis: a meta-analysis. Am Heart J. 2007 Nov;154(5):830-7. doi: 10.1016/j.ahj.2007.06.037. Epub 2007 Aug 20. PMID 17967586
- [Background] Pussinen PJ, Alfthan G, Jousilahti P, Paju S, Tuomilehto J. Systemic exposure to Porphyromonas gingivalis predicts incident stroke. Atherosclerosis. 2007 Jul;193(1):222-8. doi: 10.1016/j.atherosclerosis.2006.06.027. Epub 2006 Jul 26. PMID 16872615
- [Background] Reyes L, Herrera D, Kozarov E, Roldan S, Progulske-Fox A. Periodontal bacterial invasion and infection: contribution to atherosclerotic pathology. J Clin Periodontol. 2013 Apr;40 Suppl 14:S30-50. doi: 10.1111/jcpe.12079. PMID 23627333
- [Background] Pessi T, Karhunen V, Karjalainen PP, Ylitalo A, Airaksinen JK, Niemi M, Pietila M, Lounatmaa K, Haapaniemi T, Lehtimaki T, Laaksonen R, Karhunen PJ, Mikkelsson J. Bacterial signatures in thrombus aspirates of patients with myocardial infarction. Circulation. 2013 Mar 19;127(11):1219-28, e1-6. doi: 10.1161/CIRCULATIONAHA.112.001254. Epub 2013 Feb 15. PMID 23418311
- [Background] Offenbacher S, Beck JD, Moss K, Mendoza L, Paquette DW, Barrow DA, Couper DJ, Stewart DD, Falkner KL, Graham SP, Grossi S, Gunsolley JC, Madden T, Maupome G, Trevisan M, Van Dyke TE, Genco RJ. Results from the Periodontitis and Vascular Events (PAVE) Study: a pilot multicentered, randomized, controlled trial to study effects of periodontal therapy in a secondary prevention model of cardiovascular disease. J Periodontol. 2009 Feb;80(2):190-201. doi: 10.1902/jop.2009.080007. PMID 19186958
- [Background] Teague HL, Ahlman MA, Alavi A, Wagner DD, Lichtman AH, Nahrendorf M, Swirski FK, Nestle F, Gelfand JM, Kaplan MJ, Grinspoon S, Ridker PM, Newby DE, Tawakol A, Fayad ZA, Mehta NN. Unraveling Vascular Inflammation: From Immunology to Imaging. J Am Coll Cardiol. 2017 Sep 12;70(11):1403-1412. doi: 10.1016/j.jacc.2017.07.750. PMID 28882238
- [Background] Subramanian S, Emami H, Vucic E, Singh P, Vijayakumar J, Fifer KM, Alon A, Shankar SS, Farkouh M, Rudd JHF, Fayad ZA, Van Dyke TE, Tawakol A. High-dose atorvastatin reduces periodontal inflammation: a novel pleiotropic effect of statins. J Am Coll Cardiol. 2013 Dec 24;62(25):2382-2391. doi: 10.1016/j.jacc.2013.08.1627. Epub 2013 Sep 24. PMID 24070911
- [Background] Salminen A, Gursoy UK, Paju S, Hyvarinen K, Mantyla P, Buhlin K, Kononen E, Nieminen MS, Sorsa T, Sinisalo J, Pussinen PJ. Salivary biomarkers of bacterial burden, inflammatory response, and tissue destruction in periodontitis. J Clin Periodontol. 2014 May;41(5):442-50. doi: 10.1111/jcpe.12234. Epub 2014 Feb 17. PMID 24460823
- [Background] Meuric V, Le Gall-David S, Boyer E, Acuna-Amador L, Martin B, Fong SB, Barloy-Hubler F, Bonnaure-Mallet M. Signature of Microbial Dysbiosis in Periodontitis. Appl Environ Microbiol. 2017 Jun 30;83(14):e00462-17. doi: 10.1128/AEM.00462-17. Print 2017 Jul 15. PMID 28476771
- [Background] Bucerius J, Hyafil F, Verberne HJ, Slart RH, Lindner O, Sciagra R, Agostini D, Ubleis C, Gimelli A, Hacker M; Cardiovascular Committee of the European Association of Nuclear Medicine (EANM). Position paper of the Cardiovascular Committee of the European Association of Nuclear Medicine (EANM) on PET imaging of atherosclerosis. Eur J Nucl Med Mol Imaging. 2016 Apr;43(4):780-92. doi: 10.1007/s00259-015-3259-3. Epub 2015 Dec 17. PMID 26678270
- [Background] Rudd JH, Myers KS, Bansilal S, Machac J, Rafique A, Farkouh M, Fuster V, Fayad ZA. (18)Fluorodeoxyglucose positron emission tomography imaging of atherosclerotic plaque inflammation is highly reproducible: implications for atherosclerosis therapy trials. J Am Coll Cardiol. 2007 Aug 28;50(9):892-6. doi: 10.1016/j.jacc.2007.05.024. Epub 2007 Aug 13. PMID 17719477
- [Background] Boellaard R, Delgado-Bolton R, Oyen WJ, Giammarile F, Tatsch K, Eschner W, Verzijlbergen FJ, Barrington SF, Pike LC, Weber WA, Stroobants S, Delbeke D, Donohoe KJ, Holbrook S, Graham MM, Testanera G, Hoekstra OS, Zijlstra J, Visser E, Hoekstra CJ, Pruim J, Willemsen A, Arends B, Kotzerke J, Bockisch A, Beyer T, Chiti A, Krause BJ; European Association of Nuclear Medicine (EANM). FDG PET/CT: EANM procedure guidelines for tumour imaging: version 2.0. Eur J Nucl Med Mol Imaging. 2015 Feb;42(2):328-54. doi: 10.1007/s00259-014-2961-x. Epub 2014 Dec 2. PMID 25452219
- [Background] Bucerius J, Mani V, Moncrieff C, Rudd JH, Machac J, Fuster V, Farkouh ME, Fayad ZA. Impact of noninsulin-dependent type 2 diabetes on carotid wall 18F-fluorodeoxyglucose positron emission tomography uptake. J Am Coll Cardiol. 2012 Jun 5;59(23):2080-8. doi: 10.1016/j.jacc.2011.11.069. PMID 22651864